CLINICAL TRIAL: NCT00136409
Title: A Phase II Study of Gleevec (Imatinib Mesylate) In Patients With BCR-Negative Myeloproliferative Disorders Including Patients With Idiopathic Myelofibrosis With Myeloid Dysplasia or Chronic Myelomonocytic Leukemia
Brief Title: A Study of Gleevec in Patients With Idiopathic Myelofibrosis or Chronic Myelomonocytic Leukemia (CMML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Novartis (Industry)
Responsible Party: Principal Investigator, Daniel J. DeAngelo, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-214
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Myelofibrosis; Myeloid Metaplasia; Agnogenic Myeloid Metaplasia; Chronic Myelomonocytic Leukemia
Keywords: myelofibrosis; agnogenic myeloid metaplasia with myelofibrosis; CMML; chronic myelomonocytic leukemia; imatinib mesylate; Gleevec
MeSH Terms: conditions — Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mono-Therapy Gleevec (Experimental): Gleevec administered orally at a pre-determined dose once daily.
  Interventions: Drug: Imatinib mesylate

INTERVENTIONS:
Drug: Imatinib mesylate — 400mg orally once daily until disease progression or unacceptable side effects
  Other Names: Gleevec

SUMMARY:
The purpose of this study is to determine the effects (good and bad) of Gleevec in patients with BCR-negative myeloproliferative disorders including myelofibrosis with myeloid metaplasia and chronic myelomonocytic leukemia.

DETAILED DESCRIPTION:
Gleevec will be administered at a dose of 400 mg orally once daily.

Patients will continue to receive the drug until either drug progression or the development of intolerable side effects.

Patients will be assessed with a complete blood count weekly for the first 8 weeks and will have monthly physical examinations and bone marrow examinations every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a clinical diagnosis of myelofibrosis with myeloid metaplasia or chronic myelomonocytic leukemia (CMML). Patients may be entered based on a prior cytogenetic karyotype showing the absence of the Philadelphia chromosome.
* Patients may be entered prior to completion of reverse transcription-polymerase chain reaction (RT-PCR) or fluorescent in situ hybridization (FISH) studies, but a patient who is subsequently found to be BCR-ABL or FISH positive will be removed from protocol treatment. FISH will only be performed on patients with a normal karyotype. A PCR sample will be sent on all patients.
* The patients with myelodysplasia must have French-American-British (FAB) subtype chronic myelomonocytic leukemia (CMML) defined as peripheral blood monocytosis, and less than 30 percent blasts in the peripheral blood or the bone marrow.
* The patients with myelofibrosis with myeloid metaplasia can have one of the following: agnogenic myeloid metaplasia (idiopathic myelofibrosis), or post-polycythemic myeloid metaplasia (post-polycythemic myelofibrosis), or post-thrombocythemic myeloid metaplasia.
* Estimated life expectancy of 6 months or greater.
* Serum bilirubin equal to or less than twice the upper limit of normal.
* Serum SGOT and SGPT equal to or less than twice the upper limit of normal.
* Serum creatinine equal to or less than twice the upper limit of normal.
* Age at least 18 years.
* Greater than 4 weeks from any chemotherapy (except hydroxyurea), radiotherapy, immunotherapy, or systemic glucocorticoid therapy (non-glucocorticoid hormonal therapy is allowed). Systemic glucocorticoid therapy for non-malignant disease is allowed.
* The last dose of hydroxyurea must be 24 hours prior to the initiation of Gleevec.
* Greater than 2 months following bone marrow or peripheral blood stem cell transplantation or treatment with donor lymphocyte infusion (DLI).

Exclusion Criteria:

* Uncontrolled active infection.
* Pregnancy or nursing mothers.
* Patients with myelofibrosis with myeloid metaplasia or chronic myelomonocytic leukemia who have transformed to acute myelogenous leukemia.
* Prior treatment or diagnosis of acute myelogenous leukemia.
* Patients with Philadelphia positive cytogenetics by either peripheral blood or bone marrow sampling.
* Eastern Cooperative Oncology Group (ECOG) performance status > 3.
* Prior exposure to Gleevec.
* Active central nervous system (CNS) disease.
* Evidence of infection with the human immunodeficiency virus.
* Active psychiatric or mental illness making informed consent or careful clinical follow-up unlikely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2002-05; Primary Completion 2005-08 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To determine the overall response rate of Gleevec as a single agent in patients with BCR-negative myeloproliferative disorders including myelofibrosis with myeloid metaplasia and chronic myelomonocytic leukemia | 3 years

SECONDARY OUTCOMES:
To determine the safety and efficacy of Gleevec as a single agent in patients with BCR-negative myeloproliferative disorders including myelofibrosis with myeloid metaplasia or chronic myelomonocytic leukemia | 3 years
to determine the biologic activity of Gleevec in patients with BCR-negative myeloproliferative disorders including myelofibrosis with myeloid metaplasia or chronic myelomonocytic leukemia | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. DeAngelo, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts